CLINICAL TRIAL: NCT06131762
Title: Comparative Effects of Active and Positional Release Technique on Pain, Function and Temporospatial Gait Parameters in Runners With Plantar Fasciitis
Brief Title: Effects of Active and PRT on Pain, Function and Temporospatial Gait Parameters in Runners With Plantar Fascitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0432
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Gait; Pain; Plantar Fascitis
Keywords: pain; functions
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized control trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the reading is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active release technique (Experimental): ART performed from long sitting position, the therapist started by shortening the muscle or fascia of affected limb then apply very specific pressure with hand as we stretch tissue is lengthened. Active movement is done whenever possible according to the instructions given by therapist. ART for 8-10 minutes will be given.
  Interventions: Other: Active release technique
- Positional release technique (Experimental): Positional release technique where participant lie supine with the affected limb out of the plinth and then by application of brief mechanical pressure on tender point with one fingertip in order to determine tenderness. The foot should then be positioned, most probably into pure plantarflexion and gentle fine-tuned by rotation, until the score in the tender point has reduce by at least 70%. This position is held for 90 seconds with 3 repetitions i.e. total of 270 seconds was given.
  Interventions: Other: Positional release technique

INTERVENTIONS:
Other: Active release technique — This include active release technique for 4 weeks
  Arms: Active release technique
Other: Positional release technique — This include positional release technique for 4 weeks
  Arms: Positional release technique

SUMMARY:
The study is randomized and single -blinded. Ethical approval is taken from ethical committee of Riphah International university Lahore.Participants who will meet criteria will be requested to give verbal consent and to sign written consent form. After signing consent form participants will be allocated to the group A and Group B by using computerized generated randomization. Group A will receive ultrasound then Active release technique while group B will receive ultrasound and Positional release technique for 4 weeks. Treatment sessions will be 12 sessions, 3 sessions per week on alternative days for 4 weeks

DETAILED DESCRIPTION:
A single blinded randomized clinical trial will be conducted on 26 subjects diagnosed for planter fasciitis from Jawad Club Faisalabad and Alfatah Sports Club, Faisalabad by looking for symptoms and tenderness at heel as mentioned in inclusion criteria and will confirmed by windlass test. Participants who will meet criteria will be requested to give verbal consent and to sign written consent form. After signing consent form participants will be allocated to the group A and Group B by using computerized generated randomization. Group A will receive ultrasound then Active release technique while group B will receive ultrasound and Positional release technique for 4 weeks. Treatment sessions will be 12 sessions, 3 sessions per week on alternative days for 4 weeks. Pain will be measured by Numerical Pain Rating Scale (NPRS), Foot and ankle disability will be assessed by Foot Function Index (FFI), while gait parameters i.e. walking speed will be measured by 4-meter walking test, and step and stride length will be evaluated by measuring tape by taking foot prints before and after the 4 weeks of treatment period. Data will be analyzed through statistical package for the social sciences (SPSS) version 22.

ELIGIBILITY:
Inclusion Criteria:

* Male runners age between 18-30 years
* Duration of running at least 6 months
* Positive windlass test
* Patients with unilateral or bilateral plantar fasciitis

Exclusion Criteria:

* Recent accidental foot or ankle injury
* Previous lower-body surgical intervention within 6 months
* Recent fractures in the lower limb (femur, tibia, fibula or foot bones) within 6 months
* Diagnosed musculoskeletal disorders (rheumatoid arthritis, calcaneal spurs)
* Diagnosed neuropathy, local and systemic neurologic disorders (including sciatica, tarsal tunnel syndrome, nerve entrapment of abductor digiti minimi and posterior tibial

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Gait parameters | pre and 4 weeks post intervention
  gait parameters will be measured by 4-meter walking test
Foot Function | pre and 4 weeks post intervention
  Foot function will be assessed by Foot Function Index (FFI),

CONTACTS AND LOCATIONS:
Overall Officials: Athar Azeem, Dpt, Principal Investigator — Investigator
Locations (1):
- Jawad club, Alfatah sports complex, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brachman A, Sobota G, Marszalek W, Pawlowski M, Juras G, Bacik B. Plantar pressure distribution and spatiotemporal gait parameters after the radial shock wave therapy in patients with chronic plantar fasciitis. J Biomech. 2020 May 22;105:109773. doi: 10.1016/j.jbiomech.2020.109773. Epub 2020 Apr 3. PMID 32279933
- [Background] Waclawski ER, Beach J, Milne A, Yacyshyn E, Dryden DM. Systematic review: plantar fasciitis and prolonged weight bearing. Occup Med (Lond). 2015 Mar;65(2):97-106. doi: 10.1093/occmed/kqu177. Epub 2015 Feb 17. PMID 25694489
- [Background] Tong KB, Furia J. Economic burden of plantar fasciitis treatment in the United States. Am J Orthop (Belle Mead NJ). 2010 May;39(5):227-31. PMID 20567740
- [Background] Thong-On S, Bovonsunthonchai S, Vachalathiti R, Intiravoranont W, Suwannarat S, Smith R. Effects of Strengthening and Stretching Exercises on the Temporospatial Gait Parameters in Patients With Plantar Fasciitis: A Randomized Controlled Trial. Ann Rehabil Med. 2019 Dec;43(6):662-676. doi: 10.5535/arm.2019.43.6.662. Epub 2019 Dec 31. PMID 31918529
- [Background] Fabrikant JM, Park TS. Plantar fasciitis (fasciosis) treatment outcome study: plantar fascia thickness measured by ultrasound and correlated with patient self-reported improvement. Foot (Edinb). 2011 Jun;21(2):79-83. doi: 10.1016/j.foot.2011.01.015. Epub 2011 Mar 12. PMID 21398108